CLINICAL TRIAL: NCT06764602
Title: Observational, Retrospective, Multicenter, Nonprofit Study on the Prevalence of Renal Involvement in Pediatric Patients With Tuberous Sclerosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TSC-PED-2021-01
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Tuberous Sclerosis Complex (TSC)
Keywords: Tuberous Sclerosis Complex; Nephropathy; Children
MeSH Terms: conditions — Tuberous Sclerosis; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, retrospective, multicenter, nonprofit study on the prevalence of renal involvement in pediatric patients with tuberous sclerosis.

DETAILED DESCRIPTION:
Tuberous sclerosis (TSC) is an autosomal dominant transmission neurocutaneous syndrome caused by mutations in the TSC1 (9q34) and TSC2 (16p13.3) genes. Renal involvement in tuberous sclerosis is frequent and consists of the presence of angiomyolipomas, cysts, increased risk of renal carcinoma (predominantly clear cell renal cell carcinoma), and proteinuria in the absence of angiomyolipomas or cysts, which may evolve into chronic kidney disease. Renal involvement in tuberous sclerosis is often asymptomatic, and in most cases the finding of angiomyolipomas, cysts, or changes in renal function is an occasional finding on examinations performed during follow-up. Angiomyolipomas are the most frequent form of renal involvement in tuberous sclerosis and, when symptomatic, cause potentially fatal hemorrhages (intratumoral or retroperitoneal), anemia, hypertension, hematuria, and renal failure due to subversion of the renal parenchyma.

The renal picture of TSC (hemorrhage, end-stage renal disease, and metastasis to renal carcinoma) is the second leading cause of death in pediatric TSC patients, after neurological, and the first in the adult population. Data regarding renal involvement in the pediatric population with TSC are scarce in the literature.

This study aims to assess the prevalence of renal involvement in pediatric TSC patients. More in detail, the primary aim is to assess the prevalence of angiomyolipomas and renal cysts in pediatric TSC patients. The secondary aims are to evaluate the correlation between genetic alteration and the presence of angiomyolipomas and renal cysts in TSC patients; to evaluate the renal outcome in terms of renal function and blood pressure in pediatric TSC patients with renal involvement; to evaluate the volume change of angiomyolipomas in pediatric patients with TSC on Everolimus therapy prescribed for neurological complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex under the age of 17 years at the time of last observation (06/30/2021);
* Patients clinically evaluated in an outpatient or inpatient setting during 01/01/2018- 30/06/2021 with a diagnosis of TSC;
* Informed consent signed by parent or legal guardian.

Exclusion Criteria:

* Patients older than 18 years of age;
* Patients with other phacomatoses.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Since this is a descriptive study, a formal calculation of sample size is not expected. However, about 40-80 subjects are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Stage of angiomyolipoma | at baseline
  0-6

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pasini, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy